CLINICAL TRIAL: NCT06969378
Title: Empiric Pulsed Field Pulmonary Vein Isolation During Atrial Tachycardia Ablation in Adults With Congenital Heart Disease
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Collaborators: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Edward O'Leary, Physician, Boston Children's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-P00049906
Record Dates: First submitted 2025-05-05; First posted 2025-05-13 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Atrial Fibrillation; Atrial Tachycardia; Atrial Flutter; Congenital Heart Disease; Pulmonary Vein Isolation; Pulsed Field Ablation; Catheter Ablation
Keywords: atrial fibrillation; atrial tachycardia; atrial flutter; pulsed field ablation; congenital heart disease; adult congenital heart disease; pulmonary vein isolation; catheter ablation
MeSH Terms: conditions — Atrial Fibrillation; Atrial Flutter; Heart Defects, Congenital

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Empiric pulsed field pulmonary vein isolation (Experimental): Patients will receive general endotracheal anesthesia or conscious sedation provided by cardiac anesthesiology and usual vascular access for their clinically indicated catheter ablation for AT. Usual diagnostic methods including programmed electrical stimulation for arrhythmia induction and electroanatomic activation and voltage mapping will be performed followed by RFA (using standard-of-care, commercially-available RFA catheters) of any observed AT. After conclusion of AT ablation, transseptal or transbaffle puncture will be performed under fluoroscopic and intracardiac echocardiography guidance to access the left atrium (LA) or pulmonary venous atrium (PVA) if not already done so. PFA will be performed using a pentaspline catheter (Farawave, Boston Scientific) and a steerable sheath to achieve PVI of all veins draining to the LA/PVA with entrance and exit block confirmed at each vein. In patients where PFA is unable to achieve PVI, touch-up RFA will be performed.
  Interventions: Device: Pulsed field ablation using a pentaspline ablation catheter

INTERVENTIONS:
Device: Pulsed field ablation using a pentaspline ablation catheter — After conclusion of AT ablation, transseptal or transbaffle puncture will be performed under fluoroscopic and intracardiac echocardiography guidance to access the left atrium (LA) or pulmonary venous atrium (PVA) if not already done so. PFA will be performed using a pentaspline catheter (Farawave, Boston Scientific) and a steerable sheath to achieve PVI of all veins draining to the LA/PVA with entrance and exit block confirmed at each vein. In patients where PFA is unable to achieve PVI, touch-up RFA will be performed. Programmed atrial stimulation will be performed to investigate for inducible atrial tachycardias. An implantable loop recorder will be placed at the conclusion of the procedure.

SUMMARY:
This is a prospective, single-arm intervention trial whereby we will test the safety and efficacy of performing pulmonary vein isolation (PVI) using pulsed field ablation (PFA) in adult patients with congenital heart disease (CHD) who are presenting for atrial tachycardia (AT) ablation.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (>= 18 years of age) with repaired or unrepaired congenital heart disease and a history of sustained (>30 seconds) AT

Exclusion Criteria:

* History of sustained AF and/or previous catheter or surgical pulmonary vein isolation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Acute pulmonary vein isolation | Acute (immediate intraoperative).
  Achievement of entrance and exit block to and from all pulmonary veins draining to the left or pulmonary venous atrium.
Time to atrial tachycardia or atrial fibrillation recurrence | 12 months
  Time to sustained atrial tachycardia (AT) or atrial fibrillation (AF) lasting 30 seconds or more after a 2 month blanking period.
Major adverse event | 1 month
  Composite of stroke, transient ischemic attack, cardiac tamponade requiring percutaneous drainage, phrenic nerve injury >24 hours, atrioesophageal fistula, pulmonary vein stenosis, and/or any bleeding complication requiring blood transfusion.

SECONDARY OUTCOMES:
AT/AF Burden | 12 months
  Daily burden (measured in hours) of AT/AF as measured on an implantable loop recorder after a 2 month blanking period.
Left atrial/pulmonary venous atrial dwell time | Acute (immediate intraoperative)
  Time with sheath/catheter in left atrium or pulmonary venous atrium.
Case duration | Acute (immediate intraoperative).
  Total procedural duration (minutes)

IPD SHARING:
Plan to Share IPD: No